CLINICAL TRIAL: NCT06593236
Title: Association of Digital Aid Use With Infant Sleep and Maternal Mental Health
Status: Active, not recruiting | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Huckleberry Labs, Inc. (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nisha Fahey, Assistant Professor, University of Massachusetts, Worcester
Other Study IDs: 20242782; 1U54HL143541 (NIH)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Infant Development; Maternal Behavior
Keywords: Infant Sleep; Maternal Mental Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to better understand the use of the Huckleberry app, a pediatric sleep guidance app and the impacts on infant sleep and maternal mental health.

DETAILED DESCRIPTION:
This study aims to understand the impact of the Huckleberry app, a scalable low-cost solution to problematic child sleep patterns, on pediatric sleep and maternal mental health, especially in the Medicaid population.

A secondary aim for this study is to determine if Medicaid Accountable Care Organizations (ACO) goals are improved according to stakeholder interviews.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years old
* Has a child between the age of 0-12 months
* Receives healthcare through UMass Memorial Health
* Is a part of the Medicaid Accountable Care Organizations (ACO) population

Exclusion Criteria:

* Lacks capacity to consent
* Does not understand English
* Does not have internet access on their smartphone or at home
* If the infant is in Department of Children and Families (DCF) custody or is admitted into the Neonatal Intensive Care Unit (NICU)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will receive healthcare in the UMass Memorial Health System and must be a part of the Medicaid Accountable Care Organizations (ACO). Participants will be a birthing parent of a child aged 0-12 months.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Infant sleep quality | Baseline and 3 months
  Infant sleep quality will be assessed using the Brief Infant Sleep Questionnaire (BISQ) and will measure the quality and frequency of infant sleep. The BISQ will be delivered to participants at the baseline and endpoint of enrollment.
Maternal mental health | Baseline and 3 months
  Maternal mental health will be assessed using the Depression, Anxiety & Stress Scale (DASS21) and will assess maternal mental health. The DASS21 will be delivered to participants at the baseline and endpoint of enrollment.
Maternal bonding assessment | Baseline and 3 months
  Maternal bonding will be assessed using the Postpartum Bonding Assessment (PBQ) and will measure maternal-infant bonding. The PBQ will be delivered to participants at baseline and endpoint of enrollment.
Infant and parent sleep practices | Baseline and 3 months.
  Infant and parent sleep practices will be assessed using the Infant Sleep Practices Questionnaire. This will be a tool in assessing sleep practices. This questionnaire will be delivered to participants at baseline and endpoint of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Fahey, DO, Principal Investigator — Assistant Professor
Locations (1):
- UMass Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No